CLINICAL TRIAL: NCT00085527
Title: A Phase II Study Of Depsipeptide In Patients With Relapsed Or Refractory Ovarian Carcinoma
Brief Title: FR901228 in Treating Patients With Relapsed or Refractory Advanced Ovarian Epithelial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12965A; UCCRC-12965; LUMC-106995; NCI-6347
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Depsipeptides; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- depsipeptide (Experimental): Depsipeptide administered on Days 1, 8, and15 of a 28-day cycle.
  Interventions: Drug: depsipeptide

INTERVENTIONS:
Drug: depsipeptide
  Other Names: Romidepsin, Istodax®

SUMMARY:
RATIONALE: FR901228 may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying how well FR901228 works in treating patients with relapsed or refractory advanced ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (complete and partial) in patients with relapsed or refractory advanced ovarian epithelial carcinoma treated with FR901228 (depsipeptide).
* Determine the toxicity of this drug in these patients.

Secondary

* Correlate clinical response with platinum sensitivity in patients treated with this drug.
* Correlate clinical response with P-glycoprotein expression or p53 status in patients treated with this drug.

OUTLINE: This is multicenter study. Patients are stratified according to response to prior platinum administration (platinum resistant vs platinum sensitive).

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 20-37 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed ovarian epithelial carcinoma

  * Advanced disease
* Relapsed after OR refractory to 1, and only 1, prior platinum- or taxane-based regimen

  * Refractory disease defined as disease progression during platinum- or taxane-based therapy
  * Relapsed disease defined as platinum or taxane resistant or sensitive

    * Platinum or taxane resistance defined as relapse within 6 months after prior platinum or taxane therapy
    * Platinum or taxane sensitivity defined as relapse > 6 months from the last platinum or taxane treatment
* Measurable or evaluable disease

  * Measurable disease defined as at least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Evaluable disease determined by elevation in CA 125 (≥ 2 times upper limit of normal [ULN]), ascites, or pleural effusion
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* SWOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* At least 24 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times ULN
* Bilirubin normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* QTc < 500 msec
* LVEF > 40% by MUGA
* No significant cardiac disease
* No symptomatic congestive heart failure
* No unstable or poorly controlled angina pectoris
* No uncontrolled dysrhythmias
* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No prior serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No left ventricular hypertrophy by EKG

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Potassium ≥ 4.0 mmol/L
* Magnesium ≥ 2.0 mg/dL
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to FR901228 (depsipeptide)
* No concurrent uncontrolled illness
* No active or ongoing infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic agents

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior FR901228 (depsipeptide)
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* Prior surgical resection allowed

Other

* No concurrent drugs known to have HDI activity (e.g., sodium valproate)
* No concurrent agents that cause QTc prolongation
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent hydrochlorothiazide
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Response rate of depsipeptide in ovarian cancer | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, MD, Study Chair — University of Chicago
Locations (1):
- Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois, United States